CLINICAL TRIAL: NCT01554865
Title: The Effects of Diet-induced Weight Loss on Metabolic and Inflammatory Profile, Endothelial, Sexual and Urinary Function, and Quality of Life in Obese Men
Brief Title: Effects of Diet-induced Weight Loss in Obese Men
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2010075D
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2015-07-29 (Estimated); Status verified 2015-07

CONDITIONS: Sexual Dysfunction; Endothelial Dysfunction; Quality of Life; Inflammation
Keywords: obesity; men; sexual function; urinary tract symptoms; endothelial function; inflammation; quality of life
MeSH Terms: conditions — Sexual Dysfunction, Physiological; Inflammation; Obesity; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- conventional diet counselling (Active Comparator): counselling given by dietician on diet modification and caloric restriction
  Interventions: Behavioral: Conventional diet counseling
- partial meal replacement diet (Active Comparator): calorie-restricted diet using 1-2 meal replacements
  Interventions: Dietary Supplement: Optifast

INTERVENTIONS:
Dietary Supplement: Optifast — 1-2 sachets of Optifast daily as part of diet modification (partial meal replacement diet)
  Arms: partial meal replacement diet
Behavioral: Conventional diet counseling
  Arms: conventional diet counselling

SUMMARY:
This study aims to compare the efficacy of a partial meal replacement diet with a conventional diet, for inducing weight loss and improving metabolic and inflammatory profile, endothelial function, erectile function, sexual desire, lower urinary tract symptoms (LUTS), and quality of life in obese men.

DETAILED DESCRIPTION:
This study aims to compare the efficacy of a partial meal replacement diet with a conventional diet, for inducing weight loss, and improving metabolic and inflammatory profile, endothelial function, erectile function, sexual desire, lower urinary tract symptoms (LUTS), and quality of life in obese men. Men aged 30-65 years, with body mass index (BMI) ≥ 27.5 kg/m2, will be recruited from the community in Singapore. The study will be conducted at Changi General Hospital by trained medical investigators, dieticians and sports trainers. At baseline and 12 weeks, fasting glucose and lipids, insulin, testosterone, sex-hormone binding globulin, serum C-reactive protein and interleukin-6 are measured, endothelial function is measured by the non-invasive EndoPAT method, and validated questionnaires administered to assess changes in erectile function, sexual desire, LUTS and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 30-65 years
* Body Mass Index (BMI) >/= 27.5 kg/m2
* Waist circumference (WC) >/= 90 cm

Exclusion Criteria:

* pituitary disease or cranial radiotherapy
* previous or current androgen replacement or deprivation therapy
* current treatment for sexual problems or LUTS
* glomerular filtration rate < 60 ml/min
* liver disease
* alcohol intake exceeding 500 g/week in the previous 12 months
* use of opiates, glucocorticoids, recreational drugs or phosphodiesterase inhibitors

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
erectile function | 12 weeks
  increase in IIEF-5 score

SECONDARY OUTCOMES:
lower urinary tract symptoms | 12 weeks
  decrease in IPSS score

CONTACTS AND LOCATIONS:
Overall Officials: Joan Khoo, MBBS,MRCP, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore, Singapore